CLINICAL TRIAL: NCT04511117
Title: Endocrowns as Permanent Restorations for Endodontically Treated Permanent Molars in Young Age: Two-Year Follow up
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Roqaia Mohammad Alassar, Principal Investigator, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: PD-P-019-002
Record Dates: First submitted 2020-08-08; First posted 2020-08-13 (Actual); Last update posted 2021-12-28 (Actual); Status verified 2021-12

CONDITIONS: Endodontically Treated Teeth; Permanent Molars
Keywords: Endocrown,; Monoblock restoration,; Endodontically treated teeth; Young age
MeSH Terms: conditions — Tooth, Nonvital | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: Control group: the patient will receive direct composite resin restorations. Endocrown group: the patient will receive endocrown restorations.
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Active Comparator): ProTaper Next rotary system and iRoot SP sealer will be used for root canal treatment, followed by composite restorations.
  Interventions: Other: Control group
- Endocrown Group (Experimental): ProTaper Next rotary system and iRoot SP sealer will be used for root canal treatment, followed by endocrown restorations.
  Interventions: Other: Endocrown group

INTERVENTIONS:
Other: Control group — ProTaper Next rotary system and iRoot SP sealer with composite restorations.
  Arms: Control Group
Other: Endocrown group — ProTaper Next rotary system and iRoot SP sealer with endocrown restorations.
  Arms: Endocrown Group

SUMMARY:
Background: A real challenge faces practitioners in dealing with permanent molars in young patients starting from proper selection of endodontic treatment system till the type of final coronal restoration. For permanent molars in young age patients, which system should be followed to guarantee better performance and enhance the integrity of such weakened teeth? The question most commonly asked.

Purpose: To evaluate two-year clinical performance of endocrowns as permanent restorations for endodontically treated molars in young age.

DETAILED DESCRIPTION:
Endodontic treatment will be done for all patients using ProTaper Next rotary files and iRoot SP sealer. Then patients were randomly divided into two groups;

Gr 1: Conventional group (CG), the coronal cavity will be restored directly with bulk-fill nanohybrid composite restorations.

Gr 2: Endocrown group (EG), the coronal cavity will be restored with IPS e.max CAD endocrown restorations.

* First step: Endodontic treatment protocol will be used as the following:

  1. Biomechanical preparation using; 2.6% NaOCl for irrigation, ProTaper Next rotary files for instrumentation and 17% EDTA gel for lubrication.
  2. Obturation of root canal using; ProTaper gutta-percha and iRoot SP sealer.
* Second step: Endocrown restoration protocol will be used as the following:

  1. Occlusal Butt joint design for Endocrown preparation.
  2. Putty-wash technique for taking impression.
  3. IPS e.max CAD for Endocrown construction.
  4. G-CEM self-adhesive resin cement for Endocrown cementation.
* Follow up visits: The patients will be recalled every 6 months for evaluation.
* Evaluation methods:

  * Endodontic treatment evaluation: The outcome will be evaluated clinically and radiographically.
  * Endocrown restoration evaluation: The outcome will be evaluated clinically in terms of; marginal adaptation, marginal discoloration and surface alteration.

ELIGIBILITY:
Inclusion Criteria:

1. Patients were systemic free.
2. Mature lower permanent first molar needs conventional endodontic treatment.
3. The remaining coronal tooth structure after endodontic treatment is not less than 50%.
4. Presence of teeth in opposite arch with normal occlusion.
5. Absence of para-functional habits.
6. Supra-gingival margin after preparation.
7. No known allergies.
8. Complaint patient (parent/ guardians)

Exclusion Criteria:

1. Immature lower permanent first molar.
2. Presence of teeth, whose coronal anatomy does not allow use of rubber dam for optimum bonding.
3. Lack of cooperation of the patients to perform a postoperative radiograph and use a rubber dam for bonding.

Ages: 9 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2019-11-01 (Actual); Study Completion 2021-11-01 (Actual)

PRIMARY OUTCOMES:
Change in marginal adaptation, discoloration and surface of the restoration. | At 6 months, 12 months, 18 months, and 24 months following application.
  Alpha:
  No lack of continuity along the margin as observed with the explorer. No pigmentation anywhere on the margin.The surface of the restoration is unaltered.
  Bravo:
  Evidence of a crevice along the margin, but the explorer cannot penetrate.Pigmentation present but does not penetrate along the margin toward the pulp. The surface of the restoration shows wear, and must be controlled.
  Charlie:
  Evidence of a crevice along the margin, into which an explorer can penetrate. Requires control, repair or retreatment. Severe pigmentation. The restoration must be removed. The surface of the restoration shows perforations, fractures or significant tear. It must be polished, repaired or retreated.

SECONDARY OUTCOMES:
Change in the Retention Status. | At 6 months, 12 months, 18 months, and 24 months following application.
  Debonding or dislodgement of the restoration.

CONTACTS AND LOCATIONS:
Overall Officials: Roqaia M Alassar, DDS, Principal Investigator — Fixed Prosthodontist, Faculty of Dental Medicine for Girls, Al-Azhar University; Heba Abdelkafy, DDS, Principal Investigator — Endodontist, Faculty of Dental Medicine for Girls, Al-Azhar University; Eman Abdelraouf, DDS, Principal Investigator — Pedodontist, Faculty of Dental Medicine for Girls, Al-Azhar University
Locations (1):
- Faculty of Dental Medicine for Girls, Al-Azhar University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No